CLINICAL TRIAL: NCT04057989
Title: A Retrospective Evaluation of Ketamine Effectiveness for the Treatment of Acute Battlefield Related Pain
Brief Title: Retrospective Evaluation of Ketamine Effectiveness for the Treatment of Acute Battlefield Related Pain
Status: Completed | Type: Observational
Sponsor: Defense and Veterans Center for Integrative Pain Management (Other)
Responsible Party: Sponsor
Other Study IDs: 399623
Record Dates: First submitted 2019-08-12; First posted 2019-08-15 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Pain, Acute; Analgesia; Amputation, Traumatic; Post Traumatic Stress Disorder; Trauma, Brain
Keywords: battlefield injury; ketamine infusion; regional anesthesia; opioids
MeSH Terms: conditions — Acute Pain; Agnosia; Amputation, Traumatic; Stress Disorders, Post-Traumatic; Brain Injuries, Traumatic | interventions — Ketamine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Battlefield Injury with ketamine treatment: Patients who received ketamine infusions to treat pain from January 2007 to December 2013.
  Interventions: Drug: ketamine

INTERVENTIONS:
Drug: ketamine

SUMMARY:
Using a retrospective review of records, we will conduct a multivariate analysis to examine the relationship between exposure to ketamine, as an analgesic agent in combat related trauma care, the use of additional opioid pain medications, and patient reported pain levels.

DETAILED DESCRIPTION:
This is a retrospective study to determine if there is a relationship between intravenous infusion of ketamine given for analgesia and the use of additional opioid pain medications and patient reported pain levels before and during ketamine usage. The investigator anticipates that records of up to 700 subjects will be reviewed for eligibility. The time period 24 hours before the initial ketamine therapy is initiated along with 24 & 48 hours after the start of ketamine therapy will be the time periods examined. The average/minimum/maximum pain scores during these time periods will be used. Medication usage will be calculated over the 24 hour time periods.

This protocol is presented as an initial step in exploring the possible relationship between the administration of ketamine as an analgesic agent, the potential reduction in pain medications, and the potential reduction of pain levels. With this the goals/objectives are as follows:

Objectives

1. To compare morphine consumption in battlefield injured patients with acute pain 24 hours before the initiation of a ketamine infusion to the subsequent 48 hours following the start of infusion.
2. To compare average/minimum/maximum pain scores in battlefield injured patients with acute pain 24 hours before the initiation of a ketamine infusion to the subsequent 48 hours following the start of infusion.
3. To describe the pain trajectory in battlefield injured patients with acute pain after the initiation of ketamine infusions.
4. To measure the absolute and proportional incidence of ketamine associated side effects in battlefield injured patients with acute pain following the initiation of ketamine infusions.

ELIGIBILITY:
Inclusion Criteria:

* Battlefield injured from January 2007 to December 2013
* Prescribed a ketamine infusion for acute pain
* Awake, alert (non intubated/sedated), and able to report pain scores 24 hours prior to the start of infusion and up to 48 hours following infusion

Exclusion Criteria:

* Patients who did not receive an injury in theater and did not receive ketamine while being treated by the APS or WRNMMC/WRAMC hospital staff
* No continuous perineural catheter or epidural placement while on ketamine infusion
* Less than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female military health care beneficiaries age 18 years and older
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2014-08; Primary Completion 2017-08 (Actual); Study Completion 2017-08-30 (Actual)

PRIMARY OUTCOMES:
Opioid consumption measured in morphine equivalents | 24 hours before ketamine infusion
  Amount of opioids consumed within time frame
Opioid consumption measured in morphine equivalents | 24 hours after ketamine infusion
  Amount of opioids consumed within time frame
Opioid consumption measured in morphine equivalents | 48 hours after ketamine infusion
  Amount of opioids consumed within time frame
Pain scores | 24 hours before ketamine infusion
  Defense and Veterans Pain Rating Scale Pain scores recorded based on the Defense and Veterans Pain Rating Scale
  Rate the severity of your CURRENT pain:
  0 - No Pain
  1. - Hardly notice pain
  2. - Notice pain, does not interfere with activities
  3. - Sometimes distracts me
  4. - Distracts me, can do usual activities
  5. - Interrupts some activities
  6. - Hard to ignore, avoid usual activities
  7. - Focus of attention, prevents doing daily activities
  8. - Awful, hard to do anything
  9. - Can't bear pain, unable to do anything
  10. - As bad as it could be, nothing else matters
  Circle the number that describes how, during the past 24 hours, pain has interfered with your usual activity:
  0 - 10 (0=does not interfere, 10=completely interferes)
  Circle the number that describes how, during the past 24 hours, pain has interfered with sleep:
  0 - 10 (0=does not interfere, 10=completely interferes) Circle the number that describes how, during the past 24 hours, pain has affected your mood: 0-10
Pain scores | 24 hours after ketamine infusion
  Defense and Veterans Pain Rating Scale Pain scores recorded based on the Defense and Veterans Pain Rating Scale
  Rate the severity of your CURRENT pain:
  0 - No Pain
  1. - Hardly notice pain
  2. - Notice pain, does not interfere with activities
  3. - Sometimes distracts me
  4. - Distracts me, can do usual activities
  5. - Interrupts some activities
  6. - Hard to ignore, avoid usual activities
  7. - Focus of attention, prevents doing daily activities
  8. - Awful, hard to do anything
  9. - Can't bear pain, unable to do anything
  10. - As bad as it could be, nothing else matters
  Circle the number that describes how, during the past 24 hours, pain has interfered with your usual activity:
  0 - 10 (0=does not interfere, 10=completely interferes)
  Circle the number that describes how, during the past 24 hours, pain has interfered with sleep:
  0 - 10 (0=does not interfere, 10=completely interferes) Circle the number that describes how, during the past 24 hours, pain has affected your mood: 0-10
Pain scores | 48 hours after ketamine infusion
  Defense and Veterans Pain Rating Scale Pain scores recorded based on the Defense and Veterans Pain Rating Scale
  Rate the severity of your CURRENT pain:
  0 - No Pain
  1. - Hardly notice pain
  2. - Notice pain, does not interfere with activities
  3. - Sometimes distracts me
  4. - Distracts me, can do usual activities
  5. - Interrupts some activities
  6. - Hard to ignore, avoid usual activities
  7. - Focus of attention, prevents doing daily activities
  8. - Awful, hard to do anything
  9. - Can't bear pain, unable to do anything
  10. - As bad as it could be, nothing else matters
  Circle the number that describes how, during the past 24 hours, pain has interfered with your usual activity:
  0 - 10 (0=does not interfere, 10=completely interferes)
  Circle the number that describes how, during the past 24 hours, pain has interfered with sleep:
  0 - 10 (0=does not interfere, 10=completely interferes) Circle the number that describes how, during the past 24 hours, pain has affected your mood: 0-10
Number of ketamine side effects | 24 hours before ketamine infusion
  Recorded side effects after ketamine infusion
Number of ketamine side effects | 24 after ketamine infusion
  Recorded side effects after ketamine infusion
Number of ketamine side effects | 48 hours after ketamine infusion
  Recorded side effects after ketamine infusion

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kent, MD, Principal Investigator — Walter Reed National Military Medical Center
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States